CLINICAL TRIAL: NCT00298974
Title: A Phase 3, Randomized, Multicenter, Double-blind Study Comparing the Analgesic Efficacy of Extended Release Hydrocodone/Acetaminophen Tablets (Vicodin CR) to Placebo in Subjects With Osteoarthritis
Brief Title: A Study of Pain Relief in Osteoarthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Earle Lockhart,MD, Abbott
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M04-697
Record Dates: First submitted 2006-03-02; First posted 2006-03-06 (Estimated); Last update posted 2011-01-25 (Estimated); Status verified 2011-01

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis of the hip or knee
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Hip | interventions — Hydrocodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- hydrocodone/acetaminophen extended release (Experimental)
  Interventions: Drug: hydrocodone / acetaminophen extended release
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: hydrocodone / acetaminophen extended release — 2 tablets twice daily
  Other Names: ABT-712
  Arms: hydrocodone/acetaminophen extended release
Drug: Placebo — 2 tablets twice daily
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare the safety and pain-relieving ability of Vicodin CR to placebo in subjects with osteoarthritis (OA) of the hip or knee.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ages 21 to 80
* If female, must be of non-child bearing potential or practicing birth control
* Has osteoarthritis of the hip or knee
* Requires therapeutic doses of medication for osteoarthritis pain
* Has sufficient pain to justify the use of around-the-clock opioids

Exclusion Criteria:

* Is associated with any currently ongoing research study, or has previously participated in a Vicodin CR study
* Is allergic to or has had a serious reaction to hydrocodone, other opioids, or acetaminophen
* Cannot discontinue pain medications, even for the short time prior to the study start
* Has any clinically significant illness or recent injury, or has any significant laboratory abnormality, or has recently had major surgery
* Has a history of gastric bypass surgery or preexisting severe gastrointestinal narrowing, or history of diseases that may narrow the gastrointestinal tract
* Has a history of malnutrition or starvation
* Has a history of drug (licit or illicit) or alcohol abuse or addiction, or consumes more than 4 alcoholic drinks per day
* Has a history of a major depressive episode within the past 2 years, or requires treatment with certain drugs for depression, or has a history of major psychiatric disorder
* Pregnant or breastfeeding females
* Is incapacitated, bedridden or confined to a wheelchair
* Has initiated any new therapy or medication for OA within 1 month of screening
* Has had surgery, certain types of procedures, or received certain medications for osteoarthritis within a specified time frame
* Has other conditions that may cause pain, such as rheumatoid arthritis or gout

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 873 (Actual)
Dates: Start 2006-02; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | 12 weeks
  Arthritis Pain Intensity measured by a 100mm Visual Analog Scale (VAS)

SECONDARY OUTCOMES:
Pain intensity difference (PID) from baseline to each scheduled evaluation | 12 weeks
Western Ontario and McMaster (WOMAC) Osteoarthritis Index total score | 12 weeks
SF-36v2 Health Status Survey | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rita Jain, M.D., Study Director — Abbott
Locations (83):
- United States (83):
  - Site Ref # / Investigator 423, Birmingham, Alabama
  - Site Ref # / Investigator 581, Birmingham, Alabama
  - Site Ref # / Investigator 459, Birmingham, Alabama
  - Site Ref # / Investigator 580, Mobile, Alabama
  - Site Ref # / Investigator 479, Phoenix, Arizona
  - Site Ref # / Investigator 543, Phoenix, Arizona
  - Site Ref # / Investigator 2582, Phoenix, Arizona
  - Site Ref # / Investigator 2421, Sierra Vista, Arizona
  - Site Ref # / Investigator 453, Tempe, Arizona
  - Site Ref # / Investigator 584, Tucson, Arizona
  - Site Ref # / Investigator 393, Tucson, Arizona
  - Site Ref # / Investigator 526, Anaheim, California
  - Site Ref # / Investigator 533, Buena Park, California
  - Site Ref # / Investigator 357, Fair Oaks, California
  - Site Ref # / Investigator 721, Los Angeles, California
  - Site Ref # / Investigator 439, San Diego, California
  - Site Ref # / Investigator 709, Littleton, Colorado
  - Site Ref # / Investigator 583, Wheat Ridge, Colorado
  - Site Ref # / Investigator 497, Clearwater, Florida
  - Site Ref # / Investigator 417, Daytona Beach, Florida
  - Site Ref # / Investigator 505, DeLand, Florida
  - Site Ref # / Investigator 366, Jupiter, Florida
  - Site Ref # / Investigator 388, Longwood, Florida
  - Site Ref # / Investigator 474, Miami, Florida
  - Site Ref # / Investigator 433, Ocala, Florida
  - Site Ref # / Investigator 420, Ocala, Florida
  - Site Ref # / Investigator 359, Oldsmar, Florida
  - Site Ref # / Investigator 457, Pembroke Pines, Florida
  - Site Ref # / Investigator 434, Plantation, Florida
  - Site Ref # / Investigator 489, Plantation, Florida
  - Site Ref # / Investigator 719, Port Orange, Florida
  - Site Ref # / Investigator 481, St. Petersburg, Florida
  - Site Ref # / Investigator 2594, Tampa, Florida
  - Site Ref # / Investigator 458, West Palm Beach, Florida
  - Site Ref # / Investigator 437, Marietta, Georgia
  - Site Ref # / Investigator 2598, Meridian, Idaho
  - Site Ref # / Investigator 550, Chicago, Illinois
  - Site Ref # / Investigator 511, Evansville, Indiana
  - Site Ref # / Investigator 523, Newburgh, Indiana
  - Site Ref # / Investigator 355, Louisville, Kentucky
  - Site Ref # / Investigator 410, New Orleans, Louisiana
  - Site Ref # / Investigator 468, Owings Mills, Maryland
  - Site Ref # / Investigator 418, Pasadena, Maryland
  - Site Ref # / Investigator 560, Brockton, Massachusetts
  - Site Ref # / Investigator 715, Fall River, Massachusetts
  - Site Ref # / Investigator 522, Wellesley Hills, Massachusetts
  - Site Ref # / Investigator 527, West Yarmouth, Massachusetts
  - Site Ref # / Investigator 529, Biloxi, Mississippi
  - Site Ref # / Investigator 2544, Florissant, Missouri
  - Site Ref # / Investigator 2419, St Louis, Missouri
  - Site Ref # / Investigator 411, Omaha, Nebraska
  - Site Ref # / Investigator 389, Mamaroneck, New York
  - Site Ref # / Investigator 528, New York, New York
  - Site Ref # / Investigator 501, Roslyn, New York
  - Site Ref # / Investigator 452, Monroe, North Carolina
  - Site Ref # / Investigator 349, Winston-Salem, North Carolina
  - Site Ref # / Investigator 525, Centerville, Ohio
  - Site Ref # / Investigator 724, Cincinnati, Ohio
  - Site Ref # / Investigator 521, Cincinnati, Ohio
  - Site Ref # / Investigator 416, Cleveland, Ohio
  - Site Ref # / Investigator 582, Columbus, Ohio
  - Site Ref # / Investigator 530, Zanesville, Ohio
  - Site Ref # / Investigator 508, Oklahoma City, Oklahoma
  - Site Ref # / Investigator 723, Eugene, Oregon
  - Site Ref # / Investigator 2430, Portland, Oregon
  - Site Ref # / Investigator 493, Duncansville, Pennsylvania
  - Site Ref # / Investigator 713, Mechanicsburg, Pennsylvania
  - Site Ref # / Investigator 486, West Reading, Pennsylvania
  - Site Ref # / Investigator 351, Cranston, Rhode Island
  - Site Ref # / Investigator 466, Greenville, South Carolina
  - Site Ref # / Investigator 425, Greer, South Carolina
  - Site Ref # / Investigator 504, Milan, Tennessee
  - Site Ref # / Investigator 350, Austin, Texas
  - Site Ref # / Investigator 558, Dallas, Texas
  - Site Ref # / Investigator 727, San Antonio, Texas
  - Site Ref # / Investigator 2420, San Antonio, Texas
  - Site Ref # / Investigator 476, San Antonio, Texas
  - Site Ref # / Investigator 450, Salt Lake City, Utah
  - Site Ref # / Investigator 454, Chesapeake, Virginia
  - Site Ref # / Investigator 435, Virginia Beach, Virginia
  - Site Ref # / Investigator 556, Virginia Beach, Virginia
  - Site Ref # / Investigator 503, Virginia Beach, Virginia
  - Site Ref # / Investigator 2599, Spokane, Washington